CLINICAL TRIAL: NCT01796535
Title: An Observational, Multi Center, Non-Randomized (Single Arm) Registration of the PerX360º System™
Brief Title: The PerX360º System™ Registry
Acronym: OptiLIF™
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Interventional Spine, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TP201
Record Dates: First submitted 2012-12-10; First posted 2013-02-21 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-03

CONDITIONS: DDD

STUDY DESIGN:
Observational Model: Case-Only
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PerX360º System™: Patients treated with PerX360º System™

SUMMARY:
This is a multi-center, non-randomized post marketing surveillance registry including up to 125 patients treated with the PerX360º System™. Patients will receive a follow-up evaluation at the per physician defined time points: at discharge, an Interim 1 visit (1 month), an Interim 2 visit (3-6 months) and a Final visit (12 months). Imaging obtained at visits should be per standard of care.

DETAILED DESCRIPTION:
For all patients participating in the registry, the following outcomes will be analyzed:

* Change in pain score on the Visual Analog Scale(VAS) from baseline for leg pain
* Change in pain score on the Visual Analog Scale(VAS) from baseline for back pain
* Change in Oswestry Disability Index (ODI) score from baseline
* Proportion of patients with a device related complication
* Proportion of patients with lack of revision, removal, or reoperation
* Proportion of patients with radiographic fusion

ELIGIBILITY:
Inclusion Criteria:

* Patient understands the nature of the procedure and provides written informed consent
* Patient is willing to return to the treating physician for his/her routine follow-up visits up to 12 months post treatment
* Age > 18 years
* Patient is treated with the Optiport™ and Opticage™ products

Exclusion Criteria:None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects treated with the Optiport™ and Opticage™ products
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Fusion | 1 year
  Image Assessment

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Los Angeles Brain and Spine Institute, Los Angeles, California
  - Flagler Hospital, Saint Augustine, Florida